CLINICAL TRIAL: NCT02157610
Title: Smoking Cessation for Cervical Cancer Survivors in a Safety Net Healthcare System
Brief Title: Smoking Cessation for Cervical Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20134; R01CA172786 (NIH); NCI-2015-00067 (Registry Identifier: NCI CTRP); 2014-0204 (Other: Oklahoma University Health Services Center)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2023-04-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-02

CONDITIONS: Cervical Cancer; Tobacco Use; Smoking Cessation
Keywords: Cervical Cancer; Cervical Cancer Survivors; Smoking Cessation; Motivation And Problem-Solving; MAPS; Saliva test; Self help materials; Pamphlets; Texas Quitline; Nicotine patch; Questionnaires; Surveys; Telephone counseling sessions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Tobacco Use; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (ST) (Experimental): Participants receive free self-help materials mailed at baseline, 6, and 12 months. Participants receive a referral to the Oklahoma Quitline. Participants receive a 12-week supply of the nicotine patch and lozenge. Nicotine patch regime based on participant's self-reported smoking rate. REDCap will be used to collect all questionnaires data over the phone. Questionnaires done at baseline to randomize, then at 3, 6, 12, and 18 months. Saliva test performed at 3, 6, 12, and 18 months.
  Interventions: Behavioral: Self-Help Materials; Drug: Nicotine Patch; Behavioral: REDCap; Procedure: Saliva Test; Drug: Nicotine lozenge
- Motivation + Problem Solving (MAPS) (Experimental): Participants receive free self-help materials mailed at baseline, 6, and 12 months. Participants receive a referral to the Oklahoma Quitline.Participants receive a 12-week supply of the nicotine patch and lozenge. Nicotine patch regime based on participant's self-reported smoking rate. REDCap will be used to collect all questionnaires data over the phone. Questionnaires done at baseline to randomize, then at 3, 6, 12, and 18 months. Saliva test performed at 3, 6, 12, and 18 months. 6 telephone counseling sessions performed over 12 months. Sessions performed at baseline, 3, 6, 12, and 18 months. Sessions digitally recorded.
  Interventions: Behavioral: Self-Help Materials; Drug: Nicotine Patch; Behavioral: REDCap; Procedure: Saliva Test; Behavioral: Telephone Counseling Sessions; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Self-Help Materials — Participants receive free self-help materials mailed at baseline, 6, and 12 months. and a referral to the Oklahoma Quitline.
  Other Names: Pamphlets
Drug: Nicotine Patch — Participants receive a 12-week supply of nicotine patch. Nicotine patch regime based on participant's self-reported smoking rate. Participants who smoke >10 cigarettes/day receive 8 weeks of 21 mg, 2 week of 14 mg, and 2 week of 7 mg patches. Those who smoke <10 cigarettes/day receive 8 weeks of 14 mg and 4 weeks of 7 mg patches.
Behavioral: REDCap — REDCap will be used to collect all questionnaires data over the phone. Questionnaires done at baseline to randomize, then at 3, 6, 12, and 18 months.
  Other Names: Surveys
Procedure: Saliva Test — Saliva test performed at 3, 6, 12, and 18 months.
Behavioral: Telephone Counseling Sessions — 6 telephone counseling sessions performed over 12 months. Sessions performed at baseline, 3, 6, 12, and 18 months. Sessions digitally recorded.
  Arms: Motivation + Problem Solving (MAPS)
Drug: Nicotine lozenge — Participants receive a 12-week supply of nicotine lozenges. All participants receive 12 weeks of 2mg lozenges.

SUMMARY:
The goal of this research study is to compare a program called Motivation And Problem-Solving (MAPS) to the standard treatment to help participants with a history of cervical cancer or high-grade cervical dysplasia quit smoking.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned to 1 of 2 possible study groups. Randomization means that you are put in a group by chance, like the flip of a coin. A computer program will make this random assignment.

* If you are in Group 1, you will receive free self-help materials, and a referral to the Quitline.
* If you are in Group 2, you will receive free self-help materials, a referral to the Quitline, and 6 telephone counseling sessions over the next year. The Quitline provides free quit smoking services to eligible callers.

No matter which group you are in, you will also receive a 12-week supply of nicotine replacement therapy. The strength of the nicotine patches and lozenges you receive will depend on how much you smoke each day. You should use the nicotine patch as directed by the package instructions.

Unused and used patches have enough nicotine to poison children and pets. Be sure to fold the sticky ends together when you are done using the patch. In case of accidental overdose, call your doctor or a poison control center right away.

Even if you do not wish to use the nicotine patch, you will still be allowed to take part in the study.

Study Questionnaires:

You will be asked to complete questionnaires over the phone 5 times:

* Baseline
* Month 3
* Month 6
* Month 12
* Month 18

You will be asked about your feelings, moods, cervical cancer or dysplasia diagnosis, and smoking status. These calls should take about 45 minutes each time to complete.

Saliva Testing:

At Months 3, 6, 12 and 18, you may also be asked to provide a saliva sample to test for cotinine to confirm your smoking status. Cotinine is a chemical released in your body when it breaks down nicotine. You will receive a kit in the mail with supplies for testing. The research staff will call you to make sure that you received the kit and to discuss the instructions with you. If you have any questions about how to use the kit, you may contact the study staff during the study.

To collect the saliva, you will put a small piece of cotton in your mouth for a few minutes. You will be asked to mail the saliva sample back to the research staff, using a prepaid return envelope. You may be contacted by mail, telephone, and/or email during the study to be given reminders to send back the kit.

Telephone Counseling:

If you are in Group 2, you will have 6 telephone counseling sessions that may last up to 30 minutes each. These calls will occur over a 12-month period at times that are convenient for you. During the calls, you will be asked about how motivated you are to quit smoking, what barriers to quitting you may have, and factors that may be related to your smoking such as stress and family issues.

These sessions will be digitally recorded. The recordings will be used to help the researchers make sure that the counselors are following the correct procedures and to help the investigators better understand or improve the counseling.

Length of the Study:

Your participation in the study will end when you complete the final questionnaire call at Month 18.

If you wish to leave the study early, you should tell the study staff that you want to stop taking part in this research study. Once you tell the study staff that you want to stop participating, you will not receive follow-up questionnaire phone calls.

This is an investigational study. The nicotine patch used in this study is FDA approved and commercially available.

Up to 455 participants overall will take part in this research study.

In-Depth Interviews:

If you agree to take part in this study, you be asked to complete a questionnaire and will participate in an in-depth interview.

Demographic and Smoking History Questionnaire:

At the time of your visit you will be asked to complete a questionnaire in efforts to collect demographic and smoking history information. You may refuse to answer any question that makes you feel uncomfortable. The questionnaire may take up to 10 minutes to complete.

In-depth Interview:

You will be asked to discuss various parts of a new program designed to help women with cervical cancer quit smoking. You will be asked your thoughts on how important you think the program is, your feelings about it, and if you like it. The interview is designed to be done in a non-threatening, non-judgemental, and supportive way.

The interview should last about 2 hours.

In-depth interviews will be audio recorded and transcribed (written down).

Your participation in this study will be over when you complete the interview.

This is an investigational study.

Up to 30 women will take part in the interviews.

Up to 350 participants overall will take part in this research study. All will be enrolled at the Stephenson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Self-reported current smoker
3. History of cervical cancer or high-grade cervical dysplasia
4. Has a working telephone number
5. Has a valid home address
6. Speaks English, Spanish or both languages

Exclusion Criteria:

1. Current use of tobacco cessation medications
2. Self-report of being pregnant or lactating
3. Another household member enrolled in the study
4. Contraindication for nicotine patch use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Vidrine, PHD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma

REFERENCES:
- [Background] Vidrine JI, Sutton SK, Wetter DW, Shih YT, Ramondetta LM, Elting LS, Walker JL, Smith KM, Frank-Pearce SG, Li Y, Jones SR, Kendzor DE, Simmons VN, Vidrine DJ. Efficacy of a Smoking Cessation Intervention for Survivors of Cervical Intraepithelial Neoplasia or Cervical Cancer: A Randomized Controlled Trial. J Clin Oncol. 2023 May 20;41(15):2779-2788. doi: 10.1200/JCO.22.01228. Epub 2023 Mar 15. PMID 36921237
- [Background] Jones SR, Vidrine DJ, Wetter DW, Shih YT, Sutton SK, Ramondetta LM, Elting LS, Walker JL, Smith KM, Frank-Pearce SG, Li Y, Simmons VN, Vidrine JI. Evaluation of the Efficacy of a Smoking Cessation Intervention for Cervical Cancer Survivors and Women With High-Grade Cervical Dysplasia: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Dec 30;10(12):e34502. doi: 10.2196/34502. PMID 34967755
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment (ST): Standard Treatment (ST) consists of a mailed packet of materials including a letter referring smokers to the Oklahoma Tobacco Helpline, Florida Quitline or to the national quitline number (1-800-QUIT-NOW) for participants residing in other states, free nicotine replacement therapy when ready to quit, and standard self-help materials. ST will be mailed a total of 3 times to participants with completed assessments (Baseline, 6 and 12 months).
- Motivation + Problem Solving (MAPS): Motivation + Problem Solving (MAPS) consists of ST plus up to 6 proactive telephone counseling sessions delivered over a 12-month period. Telephone assessments across all treatment conditions will be administered at baseline and 3, 6, 12 and 18 months after baseline. The primary outcome is abstinence from tobacco at 18 months and the secondary outcomes are abstinence at other assessments, as well as quit attempts, cigarettes per day, use of the quitline across all post-baseline assessments, and cost-effectiveness.
Period: Overall Study
Arm/Group | Standard Treatment (ST) | Motivation + Problem Solving (MAPS)
Started | 100 | 102
Completed | 96 | 98
Not Completed | 4 | 4
Not completed — Death | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (ST) | Motivation + Problem Solving (MAPS) | Total
Number analyzed (Participants) | 100 | 102 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.8) | 47.5 (10.7) | 47.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 102 | 202
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 93 | 93 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 9 | 16
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 79 | 79 | 158
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 100 | 102 | 202

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Smoking Abstinence
Description: To test treatment effect at 18 months, logistic regression analysis conducted with abstinence as outcome variable, and treatment (a two-level categorical variable) as predictor, adjusting for covariates, specifically, factors used in the minimization procedures (race/ethnicity, language, age, education, income, cigarettes/day, cervical cancer stage, and time since diagnosis). A logit link and binomial variance function assumed for generalized linear mixed model (GLMM), regression and parameterize them with blocking on individual nested within treatment conditions. Treatment and time included, as well as their interaction, with adjustment for relevant covariates.
Time Frame: 18 months
Population: participants included in analysis
Measure: Number; unit: percentage
Arm/Group | Standard Treatment (ST) | Motivation + Problem Solving (MAPS)
Number analyzed (Participants) | 96 | 98
percentage | 12.9 | 14.2

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected for this project. Only all-cause mortality events were monitored during the 18 month study period.
Description: Adverse events were not collected or assessed as part of this study.
Arm/Group | Standard Treatment (ST) | Motivation + Problem Solving (MAPS)
All-Cause Mortality (participants affected / at risk) | 4/100 | 4/102
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02157610/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT02157610/ICF_000.pdf